CLINICAL TRIAL: NCT02779257
Title: Pasireotide Treatment for Insulin Producing Pancreatic Neuro-endocrine Tumor
Brief Title: Pasireotide Treatment for Neuroendocrine Tumor
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Subject passed away prior to enrollment
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Kashif Munir, Assistant Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00069513EU
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Gastro-enteropancreatic Neuroendocrine Tumor
Keywords: hypoglycemia
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Hypoglycemia | interventions — pasireotide; Diazoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pasireotide (Experimental): Off label use of pasireotide to treat refractory hypoglycemia due to an insulin-producing pancreatic neuroendocrine tumor
  Interventions: Drug: Pasireotide; Drug: Diazoxide

INTERVENTIONS:
Drug: Pasireotide — Pasireotide will be used, in addition to diazoxide, as a medical treatment to blunt hypoglycemia in the setting of autonomous insulin secretion.
Drug: Diazoxide — Pasireotide will be used, in addition to diazoxide, as a medical treatment to blunt hypoglycemia in the setting of autonomous insulin secretion.

SUMMARY:
Pasireotide binds to somatostatin receptors sst2 and sst5, which can lead to significant hyperglycemia. The investigators would like to administer pasireotide as a treatment for refractory hypoglycemia in the setting of metastatic insulin-producing pancreatic neuro-endocrine tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Biopsy-proven (primary or metastatic lesion) metastatic neuroendocrine tumor of the gastrointestinal and pancreatic location with disease determined by CT scan or MRI
3. Patients with history of clinical syndrome symptoms (e.g. hypoglycemia)
4. Patients not controlled by treatment with currently available somatostatin analogues.
5. No evidence of significant liver disease:

   * Serum bilirubin ≤1.5 x ULN
   * INR < 1.3
   * ALT and AST ≤ 3x ULN,
   * Alkaline phosphatase ≤ 2.5 x ULN
6. Written informed consent obtained prior to treatment to be consistent with local regulatory requirements
7. Is suffering from a serious or life-threatening disease or condition
8. Does not have access to a comparable or satisfactory alternative treatment (i.e., comparable or satisfactory treatment is not available or does not exist)
9. Is not eligible for participation in any of the IMP's ongoing clinical trials or has recently completed a clinical trial that has been terminated and, after considering other options (e.g., trial extensions, amendments, etc.), the clinical team has determined that treatment is necessary and there are no other feasible alternatives for the patient
10. Meets any other relevant medical criteria for compassionate use of the investigational product
11. Is not being transferred from an ongoing clinical trial for which they are still eligible
12. There are meaningful human clinical data to support an assessment that the potential benefits to patient outweigh risks.

Exclusion Criteria:

1. Patients with a known hypersensitivity to somatostatin analogs or any component of the pasireotide LAR or s.c. formulations.
2. Patients with abnormal coagulation (PT or aPTT elevated by 30% above normal limits).
3. Patients on continuous anticoagulation therapy. Patients who were on anticoagulant therapy must complete a washout period of at least 10 days and have confirmed normal coagulation parameters before study inclusion.
4. Patients currently using warfarin / warfarin derivatives
5. Patients with symptomatic cholelithiasis.
6. Patients who are not biochemically euthyroid. Patients with known history of hypothyroidism are eligible if they are on adequate and stable replacement thyroid hormone therapy for at least 3 months.
7. QT-related exclusion criteria:.

   * QTcF at screening >450 msec in males, and > 460 msec in females.
   * Family history of idiopathic sudden death
   * Sustained or clinically significant cardiac arrhythmias
   * Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block
   * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
   * Family history of long QT syndrome
   * Concomitant medications known to prolong the QT interval.
   * Potassium < or = 3.5 mmol/L
8. Patients who have any severe and/or uncontrolled medical conditions :

   * Uncontrolled diabetes as defined by HbA1c > 8%
   * Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunodeficiency, including a positive HIV test result (ELISA and Western blot). An HIV test will not be required; however, previous medical history will be reviewed.
   * Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with this study treatment.
   * Life-threatening autoimmune and ischemic disorders.
9. Patients who have a history of another primary malignancy, with the exception of locally excised non-melanoma skin cancer and carcinoma in situ of uterine cervix. Patients who have had no evidence of disease from another primary cancer for 1 or more years are allowed to participate in the study.
10. Patients with history of liver disease, such as cirrhosis or chronic active hepatitis B or C
11. Presence of Hepatitis B surface antigen (HbsAg)
12. Presence of Hepatitis C antibody (anti-HCV)
13. History of, or current alcohol misuse/abuse within the past 12 months.
14. Known gallbladder or bile duct disease, acute or chronic pancreatitis
15. Patients with hypomagnesaemia (< 0.7 mmol/L)
16. Patients with a history of non-compliance to medical regimens
17. If the patient is a sexually active male he is excluded unless he agrees to use a condom during intercourse while taking pasireotide and for 3 months after stopping pasireotide medication. They should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | up to 12 months
  number of times glucose < 70 mg/dl with and without symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kashif M Munir, MD, Principal Investigator — University of Maryland, Baltimore

REFERENCES:
- [Background] Tirosh A, Stemmer SM, Solomonov E, Elnekave E, Saeger W, Ravkin Y, Nir K, Talmor Y, Shimon I. Pasireotide for malignant insulinoma. Hormones (Athens). 2016 Apr;15(2):271-276. doi: 10.14310/horm.2002.1639. PMID 26732164